CLINICAL TRIAL: NCT03857932
Title: Clinical Study on Regularity of Lymphatic Drainage and Surgical Treatment of Breast Cancer
Brief Title: Establishment and Clinical Application of Precise SLNB System in Breast Cancer: a Randomized, Multicenter, Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qifeng Yang, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HECT004
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLNB and non-slns resection (Experimental): 1. Participants only receive SLNB
  2. preoperative CT lymphography
  3. SLNB with stained non-SLN resection
  4. SLNB with ARM dissection
  Interventions: Procedure: Participants receive SLNB as well as non SLNs resection
- SLNB group (Experimental): Participants only receive SLNB
  Interventions: Procedure: Participants receive SLNB as well as non SLNs resection

INTERVENTIONS:
Procedure: Participants receive SLNB as well as non SLNs resection — Participants only receive SLNB preoperative CT lymphography SLNB with stained non-SLN resection SLNB with ARM dissection

SUMMARY:
The investigatorsconduct the precise sentinel lymph node biopsy using preoperative computed tomographic lymphography in breast cancer. The investigators aimed to summarize the law of lymphatic drainage of breast, and to conduct the accurate surgical treatment of breast cancer.

DETAILED DESCRIPTION:
AIM:Sentinel lymph node biopsy (SLNB) is the standard technique for patients with early stage breast cancer. The investigators conduct the precise sentinel lymph node biopsy using preoperative computed tomographic lymphography in breast cancer. And The investigators identify the true sentinel lymph nodes(SLNs) followed by lymphatic ducts during operation. The investigators aimed to identify the non-sentinel lymph node, and to investigate the relationship between upper extremity lymphatic drainage. The SLNB procedure could avoid unnecessary lymph node resection and reduce treatment-related sequela.

Arm1：

1. Participants received preoperative computed tomographic lymphography
2. Participants received sentinel lymph node biopsy（SLNB）
3. Participants received stained non-sentinel lymph node resection during SLNB
4. Participants received axillary reverse mapping dissection Arm2： Participants receive sentinel lymph node biopsy

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed primary breast cancer by core needle biopsy or excisional biopsy
2. abnormal para-sentinel lymph node was found by ultrasound examination
3. ultrasound-guided fine needle aspiration cytology of these nodes were performed
4. the result of fine needle aspiration cytology was negative (no tumour cell was found)
5. participants planed to perform SLNB

Exclusion Criteria:

1. pathological diagnosed ductal carcinoma in situ by excisional biopsy
2. the result of fine needle aspiration cytology was positive
3. participants has received neo-adjuvant system therapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Up to 10 years
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to 10 years.

SECONDARY OUTCOMES:
Overall survival | Up to 10 years
  Time from randomization to death from any cause, assessed up to 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Qifeng Yang, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qifeng Yang, Jinan, Shandong, China